CLINICAL TRIAL: NCT07288710
Title: A Prospective Observational Study to Explore the Early Subjective Evaluation and Objective Recovery in Lung Cancer Patients Undergoing Sublobar Resection Versus Lobectomy
Brief Title: A Study to Explore the Early Subjective Evaluation and Objective Recovery in Lung Cancer Patients Undergoing Sublobar Resection Versus Lobectomy
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: GMU-LC-202511
Record Dates: First submitted 2025-11-19; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer (Diagnosis); Lobectomy; Sublobar Resection
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sublobar Resection Group: Patients in this group underwent sublobar resection (including segmentectomy or wedge resection). The decision for patients to receive this surgical procedure was similarly based on their routine clinical assessment, disease characteristics, physician's recommendation, and informed consent. It was not a result of randomization or active intervention by the investigators. This study will prospectively observe the post-operative recovery and prognosis of these patients, comparing them to the lobectomy group.
- Lobectomy Group: Patients in this group underwent standard lobectomy. The decision for patients to receive this surgical procedure was based on their routine clinical assessment, diagnosis, disease staging, physician's recommendation, and informed consent. It was not a result of randomization or active intervention by the investigators. This study will prospectively observe the post-operative recovery and prognosis of these patients.

SUMMARY:
The trial was designed as a single-center, non-interventional, prospective observational study to explore the role of a multimodal digital device in analyzing subjective and objective recovery in lung cancer patients undergoing sublobar resection versus lobectomy.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients (age ≥ 18 years)
2. American Society of Anesthesiologists (ASA) grade of III or below
3. scheduled for VATS from March to December 2023

Exclusion Criteria:

1. age <18 years
2. inability or poor compliance to use wearable devices
3. lack of smartphone
4. incomplete digital device data during hospitalization
5. patients with lymph node or distant metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with histopathologically confirmed lung cancer were consecutively recruited
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Electronic patient-reported outcomes | From 1 day prior to surgery through hospital discharge (assessed up to 15 days).
  The electronic patient-reported outcomes questionnaire includes pain, cough, shortness of breath, restless sleep, fatigue, drowsiness, walking difficulties, activity limitation, and distress(0 = no symptom, 10 = most severe).

SECONDARY OUTCOMES:
Length of Hospital Stay | From the day of surgery until the day of discharge, assessed up to 15 days.
  Total number of days spent in the hospital from admission to discharge.
Surgical Time | During the surgical procedure (from anesthesia induction until skin closure).
  Duration of the surgery measured in hours.
Number of Lymph Nodes Dissected | During the surgical procedure (from anesthesia induction until skin closure).
  The total count of lymph nodes harvested during the surgical procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Thoracic Surgery and Oncology, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No